CLINICAL TRIAL: NCT04552652
Title: Effect of Home-based High-Intensity Interval Training Using TeleRehabilitation Among Coronary Heart Disease Patients
Brief Title: High-intensity Interval Training and Telerehabilitation
Acronym: HIIT-TR
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: covid-19 pandemic complications with participants recruitment
Sponsor: Brno University Hospital (Other)
Responsible Party: Principal Investigator, Ladislav Batalik, Principal Investigator, Brno University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RHO58/20
Record Dates: First submitted 2020-09-11; First posted 2020-09-17 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Coronary Artery Disease
Keywords: Cardiac rehabilitatiion; Telerehabilitation; High-intensity interval training; Cardiorespiratory fitness
MeSH Terms: conditions — Coronary Artery Disease | interventions — High-Intensity Interval Training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High-intensity interval training - telerehabilitation (Experimental): 12 weeks of high-intensity interval training. Three sessions per week will be performed (36 total sessions).
  Interventions: Behavioral: High-Intensity Interval Training
- Moderate-intensity continuous training - telerehabilitation (Active Comparator): 12 weeks of moderate-intensity continuous training. Three sessions per week will be performed (36 total sessions).
  Interventions: Behavioral: Moderate-intensity continuous training

INTERVENTIONS:
Behavioral: High-Intensity Interval Training — Remotely monitored exercises will be performed at home. The high-intensity interval group warms-up for 5 minutes at moderate intensity (65-75% of maximal heart rate). After warm-up exercise, will continue in 4 minutes intervals at high-intensity to reach the target zone (85-95% of maximal heart rate) Each interval will be separated by 3 minutes of active recoveries (at 65-75% of maximal heart rate). The session ends with a 3-minute cool-down phase. Overall training exercise time will be 33 minutes - isocaloric compared to moderate-intensity continous training group. All participants will train using a heart rate monitor during each workout.
  Arms: High-intensity interval training - telerehabilitation
Behavioral: Moderate-intensity continuous training — Remotely monitored exercises will be performed at home. Patients in the moderate-intensity continuous training group will perform a 41-minute constant workout with an intensity of 65-75% of maximum heart rate, representing the same total training load as the high-intensity aerobic exercise group. All participants will train using a heart rate monitor during each workout.
  Arms: Moderate-intensity continuous training - telerehabilitation

SUMMARY:
Telerehabilitation has the potential to become an alternative attitude to outpatient cardiac rehabilitation. The aim of our study is to research the method of high-intensity interval training in the home environment using telerehabilitation. Investigators assume that the high-intensity interval training form of telerehabilitation, using a heart rate monitor as a tool for backing up training data, can improve physical fitness and lead to higher peak oxygen uptake as the traditional moderate-intensity continuous training. The study is designed as a monocentral randomized controlled trial at University Hospital Brno in the Czech Republic.

After the coronary event, eligible patients will be randomly (in 1:1 ratio) separated into two groups: the experimental high-intensity interval training group and the moderate-intensity continuous control group. Both groups undergo a 12-week telerehabilitation training program with a 52-week follow-up period. The primary outcome observed will be the effect of intervention expressed by changes in peak oxygen uptake values.

DETAILED DESCRIPTION:
The study relates to the previous study project CR-GPS, in which investigators proved the feasibility of cardiac telerehabilitation. The results showed that aerobic capacity and quality of life improved similarly in telerehabilitation and outpatient group of participating patients. During the research, investigators used the moderate-intensity continuous method. The present research focuses on high-intensity interval training, which presents comparable or even better results in cardiorespiratory condition effects and requires less time than a continuous method in patients with low or medium cardiovascular risk.

ELIGIBILITY:
Inclusion Criteria:

* Participants with coronary artery disease (in last two months)
* with low or medium cardiovascular risk
* with heart revascularization
* with recommended pharmacotherapy
* with clinically stable state
* with the ability to perform a cardiopulmonary exercise test
* with the ability to understand and write in the Czech language
* with an internet connection at home
* literacy with information and communication technology

Exclusion Criteria:

* Participants who were hospitalized with heart disease in the previous six weeks
* with psychological severe or cognitive disorders
* with contraindications for cardiopulmonary exercise testing
* with severe training limitations besides coronary artery disease
* with a planned intervention or operation
* participants who are enrolled in or participate in an outpatient form of cardiac rehabilitation
* participants who plan to be or are included in other studies

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2023-07-25 (Actual); Study Completion 2023-07-25 (Actual)

PRIMARY OUTCOMES:
Cardiorepisratory fitness (CRF) | Change from baseline to 12 weeks and 52weeks
  Peak oxygen uptake (VO2peak) during cardiopulmonary exercise test

SECONDARY OUTCOMES:
Health-related quality of life (SF-36 Form) | Change from baseline to 12 weeks and 52weeks
  The SF-36 yields a score for each domain of health. All domains are scored on a scale from 0 (negative health) to 100 (positive health), with 100 representing the best possible health state.
Hospital Anxiety and Depression scale (HADS) | Change from baseline to 12 weeks and 52weeks
  The questionnaire comprises seven questions for anxiety and seven questions for depression. Each item on the questionnaire is scored from 0-3 and this means that a person can score between 0 and 21 for either anxiety or depression.
Satisfaction - self-completed questionnaire | 12 weeks and 52weeks
  Subjects will be provided with a 5-item self-completed questionnaire developed by our research team that will measure their satisfaction with the intervention they received and the study in general. The items will be presented in the form of statements to which subjects will be asked to respond using a 1-5 Likert scale ("strongly agree", "agree", "not sure", "disagree", and strongly disagree").
Body composition (BIA) | Change from baseline to 12 weeks and 52weeks
  Total muscle mass, fat mass and body water will be measured by bioelectrical impedance analysis.
Incidence of treatment-emergent adverse events assessed by 5 grade scale | Data will be recorded continuously from the intervention's baseline for 12 weeks and then for 52 weeks.
  Participants will be encouraged to use the contact details for reporting incidence of treatment-emergent adverse events at any time throughout the study period.
  The type, incidence, and severity of adverse events by scale (Grade 1: Mild, asymptomatic or mild symptoms; Grade 2: Moderate, minimal; Grade 3: Severe or medically significant; Grade 4: Life-threatening consequences; and Grade 5: Death) will be noted.
Training adherence (Number of compliant participants, Average exercise time, Overall completition rate) | 12 weeks
  Adherence to the training will be recorded in the exercise datasheets from the telemonitoring platform.
  Evaluation of:
  * the overall completion rate of prescribed exercise lessons (100% = 36)
  * the total average time of all exercises in the defined heart rate zone
  * the total number of compliant participants (The criterium of compliance with the rehabilitation program is set at 70% of the prescribed training lessons)
Anxiety (General anxiety disorder, 7-item scale) | Change from baseline to 12 weeks and 52weeks
  Monitoring efficacy by score on a seven-item scale of generalized anxiety disorder. General anxiety disorder, 7-item scale total score for the seven items ranges from 0 to 21. 0-4: minimal anxiety. 5-9: mild anxiety. 10-14: moderate anxiety. 15-21: severe anxiety.

CONTACTS AND LOCATIONS:
Overall Officials: Filip Dosbaba, PT, PhD, Principal Investigator — University Hospital Brno, Czech Republic
Locations (1):
- University Hospital Brno, Brno, Czechia

IPD SHARING:
Plan to Share IPD: Yes
there is a plan to make the data on each participant available to other researchers through a web-based data register
Supporting Information: Study Protocol, CSR
Time Frame: 2020 - 2024
Access Criteria: unlimited, open access